CLINICAL TRIAL: NCT03889184
Title: An Innovative Rehabilitating Meals-on-wheels Service for Frail Old People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anne Marie Beck, senior associate professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DGK
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Undernutrition; Rehabilitation
Keywords: meals-on-wheels; home-dwelling older people
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rehabilitating meals-on-wheels service (Experimental): the intervention group will for 8 weeks receive a rehabilitating meals-on-wheels service
  Interventions: Other: rehabilitating meals-on-wheels service
- Usual care (No Intervention): the control group will receive usual care

INTERVENTIONS:
Other: rehabilitating meals-on-wheels service — the meals-on-wheels service will be specifically targeted for old people discharged from hospital, receiving exercise rehabilitation in the municipality or already receiving meals-on-wheels
  Arms: rehabilitating meals-on-wheels service

SUMMARY:
The aim of the project is to assess the beneficial effect of offering frail old people a targeted meals-on-wheels service in 8 weeks in a randomized controlled trial

DETAILED DESCRIPTION:
The aim of the project is to assess the beneficial effect of offering frail old people a targeted meals-on-wheels service in 8 weeks in a randomized controlled trial. The target group is, respectively old people discharged from an hospital stay, old people referred for exercise rehabilitation in the municipality and old people already receiving meals-on-wheels

ELIGIBILITY:
Inclusion Criteria:

* 65+ year,
* able to speak and understand Danish.
* has accepted to participate
* Is discharged from hospital, or
* is referred to exercise rehabilitation in the municipality or
* is receiving meals-on-wheels

Exclusion Criteria:

* terminal disease,
* living in a nursing home,
* receives a specific diet (e.g. diabetes, dysphagia, vegetarian or vegan)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
EuroQoL (EQ-5D-5l) | change after 8 weeks
  (EQ-5D-3L) is a standardized instrument for use as a measure of health outcome. The EQ-5D-5L descriptive system comprises the following 5 dimensions (5D): mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension has 5 levels (5L): from no problems (1 point), to extreme problems (5 points).
readmissions | after 30 days
  measuring prevalence of hospital admissions within 30 days
protein intake | change after 8 weeks
  assessment of dietary intake of protein by means of a 24 hour recall

SECONDARY OUTCOMES:
physical function | change after 8 weeks
  30-seconds chair stand
Satisfaction with food-related quality of life questionnaire (SWFL) | change after 8 weeks
  SWFL consist of five items that can be measured independently, or grouped into a single dimension. The participants evaluate their degree of agreement, with five statements of answer possibilities (from disagree completely to agree completely), and a higher level means a better SWFL score.
Food related functional ability questionnaire (scale) | change after 8 weeks
  Food-related functional ability is assessed based on questions of ability (or inability) to handle shopping, table coverage, cooking, heating and eating, as well as being able to chew and swallow food without problems and to see, hear, smell and taste food. There are four response categories from 'yes, effortlessly' to 'no, not at all'. In addition, six questions regarding the extent to which the participant can master daily chores regarding today's main meals. There are five response categories from "" can not at all "to" to very much ".
Meal quality questionnaire | change after 8 weeks
  meal quality is assessed on the basis of the Nutrition and Health Education's culinary assessment schedule, which includes seven assessment criteria, as well as supplementary questions about the correspondence between the citizen's expectations and the appearance of the food. The assessment criteria include sensory factors regarding the appearance of the food, fragrance, taste, consistency, temperature, portion size and overall assessment. The criteria are assessed on a Likert scale (1-5), where 1 is defined as very poor and 5 is defined very well.
Compliance | after 8 weeks
  assessment of percentage of use of provided meals-on-wheel service
adverse events | during the 8 weeks
  assessment of adverse events related to the intervention, e..g number of partiicpants with nausea,

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Beck, PhD, Principal Investigator — University College Copenhagen
Locations (1):
- Municipality of Albertslund, Albertslund, Denmark